CLINICAL TRIAL: NCT00967720
Title: Qualitative Analysis of the Barriers to Adherence With Asthma Controller Medication Among Inner City African American Adolescents as Identified Through Focus Group Data
Brief Title: Barriers to Adherence to Asthma Controller Meds in Low Income Urban Minority Adolescents
Acronym: ADEPT
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Giselle Mosnaim, MD, Rush University Medical Center
Other Study IDs: 08021601
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barriers, Adherence, Asthma

SUMMARY:
Poor adherence to appropriate asthma medications is an important risk factor contributing to high asthma morbidity and mortality in urban African American adolescents. As part of the ADEPT (Adolescent Disease Empowerment and Persistency Technology) for Asthma Pilot 2 study, a focus group was developed specifically to explore existing barriers to adherence among inner city African American adolescent asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age
* self identify as African American
* have persistent asthma
* read at a minimum fourth grade reading level
* be on a prescribed daily inhaled corticosteroid medication for asthma

Exclusion Criteria:

* candidate refusal or presence of other co-morbidities

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: four low income urban adolescents with uncontrolled moderate persistent asthma
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Focus groups explored whether a new communication medium improved adherence to asthma controller medications and to examine existing barriers to adherence among four urban African American adolescents with uncontrolled moderate persistent asthma

CONTACTS AND LOCATIONS:
Overall Officials: Giselle S Mosnaim, MD, Principal Investigator — Rush University Medical Center